CLINICAL TRIAL: NCT05466578
Title: Pre-approval Single-patient Expanded Access for Abrocitinib (PF-04965842)
Status: Available | Type: Expanded Access
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B745
Record Dates: First submitted 2022-06-22; First posted 2022-07-20 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-09

CONDITIONS: Severe Uncontrolled Atopic Dermatitis
Keywords: atopic dermatitis; AD; Atopic eczema; JAK inhibitors
MeSH Terms: conditions — Dermatitis, Atopic | interventions — abrocitinib

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: abrocitinib

SUMMARY:
Provide pre-approval single patient Expanded Access (compassionate use) of abrocitinib for patients with severe uncontrolled atopic dermatitis

DETAILED DESCRIPTION:
In Expanded Access, treating physicians are the Sponsor.

Expanded Access requests from treating physicians may be submitted at www.pfizercares.com ; availability will depend on location/country.

ELIGIBILITY:
Must have severe uncontrolled atopic dermatitis refractory to other available treatments

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult